CLINICAL TRIAL: NCT05791214
Title: Evalution of Nurse's Specific Abilities in ICU Setting: Creation and Validation of a New Score
Brief Title: Evalution of Nurse's Abilities in ICU Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Oliva Matrona, nurse, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5106
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Assessment Tool of Nurses' Skills

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: score — Creation and validation of new nurse' score in ICU

SUMMARY:
The assessment of nurses' skills is of fundamental importance in order to predict their performance, this is true in all areas of care but especially in the critical area. The aim of the single center prospective observational study is to provide the organization and specifically the nursing coordinator with an evaluation form that is as specific and complete as possible for evaluating the performance of nurses in ICU.

The nursing coordinators of 4 UOCs of intensive care for adults in the IRCCS Gemelli Polyclinic Foundation in Rome will be involved in the use of an evaluation scale for nurses. In each UOC, 10 nurses will be randomly selected for which to carry out the evaluation, subject to informed consent and compliance with the inclusion criteria in the study.

Results Certify the reliability of the Scale for evaluating the performance and attitudes of nurses working in intensive care.

It is hypothesized that an objective assessment tool of nurses' skills allows for an adequate allocation of resources not only in quantitative terms but also and above all in qualitative terms.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care nurses present for at least 12 months in the relevant unit,

Exclusion Criteria:

* Newly hired or newly transferred nurses (<12 months of presence in the relevant ICU).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The coordinator nurses of the ICU, considered collaborators of the PI, will use the Scale for the evaluation of 10 nurses belonging to their staff, as in the case of the usual annual performance evaluation, therefore only once per person
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
evaluation the performance of nurse in ICU | 2 years
  Certify the reliability of the Scale for evaluating the performance and attitudes of nurses working in intensive care.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli, Roma, Italy